CLINICAL TRIAL: NCT00301990
Title: A Phase II Study of Bevacizumab and Aldesleukin in Patients With Metastatic Renal Cell Carcinoma (RCC): A Cytokine Working Group (CWG) Study
Brief Title: Bevacizumab and Interleukin-2 in Treating Patients With Metastatic Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000460074; UCLA-050658-01; DMS-W0454; NCT00142142 (obsolete NCT alias)
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2007-04

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Bevacizumab

INTERVENTIONS:
Biological: aldesleukin
Biological: bevacizumab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Interleukin-2 may stimulate the white blood cells to kill tumor cells. Giving bevacizumab together with interleukin-2 may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with interleukin-2 works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the response, progression-free survival, and overall survival of patients with metastatic renal cell carcinoma (RCC) treated with bevacizumab and high-dose interleukin-2 (IL-2).

Secondary

* Compare the response and survival of patients with metastatic RCC treated with bevacizumab and high-dose IL-2 with the historical data of patients treated with high-dose IL-2 alone.
* Compare the toxicity of bevacizumab and high-dose IL-2 in patients with metastatic RCC with the historical data of patients treated with high-dose IL-2 alone, in terms of number of doses of IL-2 administered during the first course of therapy, toxicity after the scheduled ninth dose of IL-2, and frequency of grade III and IV or unexpected or rare toxicities.
* Compare the time to disease progression in patients with metastatic RCC treated with bevacizumab and high-dose IL-2 with the historical data of patients treated with high-dose IL-2 alone.
* Evaluate the pharmacokinetics and pharmacodynamics of bevacizumab and high-dose IL-2 during course 1.
* Correlate serum vascular endothelial growth factor (VEGF) levels, DC function, TCR zeta chain expression, and arginase or arginine levels with toxicity, response, and survival of patients treated with this regimen.
* Evaluate the utility of known prognostic criteria for RCC patients on clinical outcome.

OUTLINE: This is a multicenter study. Patients are stratified according to prognosis (good vs intermediate vs poor).

Patients receive bevacizumab IV over 30-90 minutes on days -13, 1, 15, 29, 43, 57, and 71 during course 1 and on days 1, 15, 29, 43, 57, and 71 during courses 2 and 3. Patients also receive high-dose interleukin-2 every 8 hours on days 1-5 and 15-19. Treatment repeats every 84 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell carcinoma (RCC) with predominantly clear cell histology
* Measurable disease
* No history of tumor-related hemorrhage
* No history of CNS or brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status ≥ 80%
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusion or recombinant erythropoietin growth factors allowed)
* AST ≤ 2 times upper limit of normal (ULN) (5 times ULN if due to liver metastases)
* Serum total bilirubin ≤ 2 times ULN (except for patients with Gilbert's disease)
* Serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* FEV_1 ≥ 2.0 L or ≥ 75% of predicted

  * Pulmonary function testing required for patients over age 50 or with significant pulmonary or smoking history
* No history of cerebrovascular accident or transient ischemic attacks
* No evidence of any of the following cardiac conditions*:

  * Congestive heart failure
  * Symptoms of coronary artery disease
  * Myocardial infarction < 6 months prior to study entry
  * Serious cardiac arrhythmias
  * Unstable angina NOTE: *Patients > 40 years old or who have had a previous myocardial infarction > 6 months prior to study entry are required to have a negative or low probability cardiac stress test for cardiac ischemia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except nonmelanoma skin cancer or noninvasive cancer, such as cervical carcinoma in situ, superficial bladder cancer without local recurrence, or breast cancer in situ

  * Patients with a history of another invasive malignancy must be in complete remission for ≥ 5 years
* No positive serology for HIV, hepatitis B, or hepatitis C
* No significant co-morbid illness, such as uncontrolled diabetes or active infection, that would preclude study treatment
* No history of inflammatory bowel disease or other serious autoimmune disease

  * Thyroiditis or rheumatoid arthritis allowed
* No uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg)
* Proteinuria ≤ 3+ by dipstick OR proteinuria < 2 gm by 24-hour urine collection
* Urine protein:creatinine ration < 1.0
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study entry
* No significant traumatic injury within the past 28 days
* No serious, nonhealing wound, ulcer, or bone fracture
* No active bleeding
* No history of other serious hemorrhage, bleeding diathesis, or underlying coagulopathy
* No history of deep venous thrombosis, clinically significant peripheral vascular disease, or other thrombotic event

PRIOR CONCURRENT THERAPY:

* No organ allografts
* At least 4 weeks since prior radiotherapy or surgery and recovered
* No prior systemic therapy for metastatic RCC
* No prior bevacizumab or interleukin-2
* At least 2 weeks since prior steroids
* No major surgery or open biopsy within the past 28 days
* No minor surgical procedures, fine needle aspirations, or core biopsies within the past 7 days, except central venous catheter placement
* No concurrent major surgery
* No concurrent corticosteroids or other immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2005-09

PRIMARY OUTCOMES:
Response
Progression-free and overall survival

SECONDARY OUTCOMES:
Comparison of response and survival with historical data
Toxicity
Time to disease progression
Pharmacokinetics and pharmacodynamics
Correlation of serum VEGF levels, DC function, TCR zeta chain expression, and arginase or arginine levels with toxicity, response, and survival
Utility of known prognostic criteria

CONTACTS AND LOCATIONS:
Overall Officials: Fairooz F. Kabbinavar, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (11):
- United States (11):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia